CLINICAL TRIAL: NCT03972579
Title: Behavioral Profile Matching: A Precision Medicine Approach to Concussion Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Noah Silverberg, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H18-02344
Record Dates: First submitted 2019-05-22; First posted 2019-06-03 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded exposure therapy (Active Comparator): Weekly 60-min sessions with an occupational therapist and psychologist over 8 weeks.
  Interventions: Behavioral: Graded exposure therapy
- Pacing + mindfulness (Active Comparator): Weekly 60-min sessions with an occupational therapist and psychologist over 8 weeks.
  Interventions: Behavioral: Pacing + mindfulness

INTERVENTIONS:
Behavioral: Graded exposure therapy — Gradually increased contact with avoided sensory stimuli (e.g., light, noise, movement) and activities (e.g., mental exertion, physical exercise, stressful activities) in order to increase tolerance.
  Arms: Graded exposure therapy
Behavioral: Pacing + mindfulness — Shifting from symptom-contingent to time-contingent activity stopping rules, minimizing activity level peaks (excessive endurance behavior) and valleys (prolonged periods of recuperative rest) to improve overall functioning.
  Arms: Pacing + mindfulness

SUMMARY:
At least 1 in 5 people who sustain a concussion will have persistent symptoms and difficulties with daily activities. The researchers have identified two unhelpful coping styles following a concussion - avoidance and endurance. Individuals who engage in avoidance behavior may benefit from a different type of treatment than those who engage in endurance behavior. The researchers will evaluate whether assigning individuals to a specific psychologically-informed treatment tailored to their coping style is practical, acceptable, and beneficial for their recovery.

DETAILED DESCRIPTION:
Psychosocial factors are known to affect recovery from concussion, but are not sufficiently taken into account by current treatment approaches. Distinct behavioral profiles after concussion have emerged in our research: (1) avoidance, where individuals perceive activity as overly dangerous and take care to avoid overexertion, and (2) endurance, where individuals persist with high levels of activity despite worse symptoms until they "crash," requiring recuperative rest. The researchers hypothesize that patients with these behavioral profiles likely benefit from different treatment approaches. The next step in our research program is to evaluate the feasibility and potential impact of tailoring therapies based on an Avoidance-Endurance Model adapted from the chronic pain literature.

The proposed project aims to evaluate whether matching patients with concussion to tailored therapies based on their behavioral profile (avoidance vs endurance) is feasible. A secondary aim is to test our hypothesis that participants receiving the intervention matched to their behavioral profile will have less post-treatment disability than mismatched participants.

In a pilot double-blind (patient, assessor) RCT with 1:1 allocation stratified by behavioral profile (avoidance vs. endurance), 64 adults with persistent symptoms after concussion will complete an initial evaluation, an activity diary over the following week, and then be randomized to receive an interdisciplinary treatment package tailored to avoidance or endurance profiles.

In brief, the program designed for avoidance will involve graded exposure to cognitively demanding activity (e.g., mental math exercises), physical exertion (e.g., treadmill jogging), and sensory stimulation (e.g., scenes with visual motion). The focus of the endurance program will be pacing, i.e., shifting from symptom-contingent to time-contingent behavior. A blinded assessor will administer outcome measures 12 weeks after enrollment. Feasibility criteria include acceptability of randomization and treatment tolerability, fidelity, and adherence.

Proposed changes to "profile matching" study due to COVID-19 pandemic (March 30, 2020)

Due to the COVID-19 pandemic, there will be no new enrollments as of March 30, 2020. The study will continue to be advertised at concussion clinic group education sessions, which are now being held virtually, but inform prospective participants that enrollment will be postponed by at least one month. Interested patients will be added to a waitlist for screening when the study resumes enrollment (once COVID-19 social distancing restrictions are lifted and non-essential business/services are resumed).

For participants who have expressed interest in the study and/or have already been screened, but have not completed their baseline assessment: Defer baseline assessment. Inform the participant that the study will resume enrolling when COVID-19 restrictions have been lifted. They will keep their place on a study waitlist. Patients who have been screened will need to be re-screened when enrollment resumes.

For participants who have completed their baseline assessment or are already active in treatment: Continue treatment per protocol. However, participants who have completed no more than 25% of treatment (4 of 16 sessions) should be offered the option of a temporary stoppage for at least one month (i.e., the target of completing all 16 sessions within 10 weeks can be dropped). If the therapists believe that treatment progress is being significantly impeded by COVID-19 restrictions, they may suggest a stoppage. The final decision about stoppage should be made by the participant. If they prefer a stoppage, the therapists should contact the participant in one month to decide whether to resume treatment or delay by another month. Any stoppages should be communicated to the study coordinator.

For participants who completed treatment, or at least 75% of their treatment (12 of 16 sessions), by March 13, 2020 but did not complete their outcome assessment until after that date: Complete the outcome assessment per protocol, but add one question immediately following the WHODAS. Introduce the question as follows:

"These questions were about how much difficulty you had with various activities due to your health conditions over the past month. In other words, I asked you focus on difficulties caused by your concussion and/or other health conditions. However, the investigators recognize that it might be hard to ignore circumstances other than your health conditions when answering these questions." Ask: "To what extent were your answers to these questions affected by the COVID-19 pandemic?" If they ask what "affected by the COVID-19 pandemic" means, the research assistant may provide examples: "Such as all of sudden being laid off or asked to work overtime, or not being able to go out because of social distancing policies." Provide responses: 0=minimally or not at all, 1=somewhat, 2=quite a bit, 3=very much or entirely.

Confirm their response by asking "So, were it not for the COVID-19 pandemic, would you have answered these questions ___________ differently?" Please also record (free text) notes if participants provide explanations or reasons. Note that this additional question is being asked only for the primary study outcome (WHODAS). This question will be removed from the protocol one month after COVID-19 social distancing restrictions are lifted and non-essential business/services are resumed.

Changes to the statistical analysis plan:

Participants whose treatment progress and/or outcome assessment was likely substantially impacted by COVID-19 will be excluded from the primary analysis. Participants who treatment progress and/or outcome assessment was possibly mildly impacted, but not likely substantially impacted, by COVID-19 will be included in the primary analysis. This will be operationalized according to the Table 1 below.

Participants who are eligible (completed no more than 4 therapy sessions by March 30, 2020) and choose to temporarily stop treatment during the COVID-19 disruption period will not be counted in the numerator or denominator for calculating the retention rate as a feasibility outcome.

Coding the COVID_status variable: 0

Operational definition:

0a. Participants who completed their outcome assessment by March 13, 2020. 0b. Participants who completed at least 75% of their treatment (12 of 16 sessions) by March 13, 2020 and the outcome assessment between March 14 and on April 30*, and answered 0 or 1 to the WHODAS COVID question.

0c. Participants who completed no more than 25% of their treatment (0-4 therapy sessions) by March 30, 2020 and agreed to temporarily stop treatment (before their 5th therapy session) until after April 30, 2020*.

0d. Participants who enrolled after April 30, 2020*. 0e. Participants who meet criteria 1b or 1c (below) but both of their therapists agreed with the statement "therapy goals and progress were not affected by COVID-19" and the participant answered 0 or 1 to the WHODAS COVID question.

-Represents participants whose therapy progress and outcome assessment were minimally or not affected by COVID-19 disruptions. It captures participants who did most or all of their therapy outside of the COVID-19 disruption period, as well as the few who continued therapy unimpeded by COVID-19 disruptions. These participants will be included the primary analysis.

Coding the COVID_status variable: 1

Operational definition:

1a. Participants who completed at least 75% of their treatment (12 of 16 sessions) by March 13, 2020 and their outcome assessment between March 14-April 30, 2020*, and answered 2 or 3 to the WHODAS COVID-19 question.

1b. Participants who completed more than 25% but less than 75% of their treatment (i.e., 5-11 sessions) by March 30, 2020, and do not meet criterion 0e.

1c. Participants who completed no more than 25% of their treatment (0-4) by March 30, 2020 and chose to continue treatment during the period in which COVID-19 social distancing restrictions, and do not meet criterion 0e.

-Represents participants whose therapy progress and/or outcome assessment were likely affected by COVID-19 disruptions. These participants will be excluded from primary analysis.

*Note: March 14, 2020 is the start of the COVID-19 disruption period in British Columbia, when the first social distancing policies were introduced. April 30, 2020 is a placeholder date for when COVID-19 social distancing restrictions are lifted and non-essential business/services are resumed. The actual date will be updated.

ELIGIBILITY:
Inclusion criteria:

* Aged 18-70 years old.
* Sustained a mild traumatic brain injury between 1 and 12 months ago.
* Fluent in English.
* Access to a computer, tablet, or smartphone with internet capability.
* 3+ persistent moderate-severe symptoms on the Rivermead Postconcussion Symptom Questionnaire.
* High avoidance (Fear Avoidance Behavior after Traumatic Brain Injury; FAB-TBI) and/or endurance behavior (Behavioral Response to Illness Questionnaire - All-Nothing subscale).

Exclusion criteria:

* Patients with a cardiac contraindication to aerobic exercise will be excluded

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
World Health Organization Disability Assessment Schedule (WHODAS) 2.0 12-item | Initial assessment, past 30 days.

SECONDARY OUTCOMES:
Rivermead Postconcussion Symptom Questionnaire | initial assessment, past 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Silverberg, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehab Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Shi S, Picon EL, Rioux M, Panenka WJ, Silverberg ND. Catastrophizing is associated with excess cognitive symptom reporting after mild traumatic brain injury. Neuropsychology. 2024 Feb;38(2):126-133. doi: 10.1037/neu0000930. Epub 2023 Nov 2. PMID 37917438
- [Derived] Mikolic A, Panenka WJ, Iverson GL, Cotton E, Burke MJ, Silverberg ND. Litigation, Performance Validity Testing, and Treatment Outcomes in Adults With Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2024 May-Jun 01;39(3):E153-E161. doi: 10.1097/HTR.0000000000000903. Epub 2023 Sep 29. PMID 37773600
- [Derived] Terpstra AR, Louie DR, Iverson GL, Yeates KO, Picon E, Leddy JJ, Silverberg ND. Psychological Contributions to Symptom Provocation Testing After Concussion. J Head Trauma Rehabil. 2023 Mar-Apr 01;38(2):E146-E155. doi: 10.1097/HTR.0000000000000796. Epub 2022 Jun 9. PMID 35687896
- [Derived] Silverberg ND, Cairncross M, Brasher PMA, Vranceanu AM, Snell DL, Yeates KO, Panenka WJ, Iverson GL, Debert CT, Bayley MT, Hunt C, Baker A, Burke MJ; Canadian Traumatic Brain Injury Research Consortium (CTRC). Feasibility of Concussion Rehabilitation Approaches Tailored to Psychological Coping Styles: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Aug;103(8):1565-1573.e2. doi: 10.1016/j.apmr.2021.12.005. Epub 2021 Dec 28. PMID 34971596
- [Derived] Terpstra AR, Cairncross M, Yeates KO, Vranceanu AM, Greenberg J, Hunt C, Silverberg ND. Psychological mediators of avoidance and endurance behavior after concussion. Rehabil Psychol. 2021 Nov;66(4):470-478. doi: 10.1037/rep0000390. Epub 2021 Aug 19. PMID 34410757